CLINICAL TRIAL: NCT00746434
Title: A Proof of Concept Study With 0.5% Roflumilast Cream in Patients With Mild to Moderate Plaque Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to business decisions. No subjects were treated.
Sponsor: AstraZeneca (Industry)
Collaborators: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO-2351-002-EM
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Plaque Psoriasis
Keywords: Mild plaque psoriasis,; Moderate plaque psoriasis,; 0.5% Roflumilast cream

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Roflumilast cream 0.5%
  Interventions: Drug: Roflumilast cream
- 2 (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Roflumilast cream — Roflumilast cream 0.5%
  Arms: 1
Drug: Placebo cream — Placebo cream
  Arms: 2

SUMMARY:
The aim of this proof of concept study is to show the safety and efficacy of 0.5 % dermal roflumilast cream in the treatment of plaque psoriasis in adults. This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study. 3-10 % of the body surface area (BSA) should be covered with a mild to moderate form of plaque psoriasis. In a 4-week treatment period 76 mg cream is applied two times daily on up to 2% of the BSA. After a screening phase, a washout phase of flexible duration (max 30 days, time depending upon pre-medication), the 28 day treatment phase follows. As roflumilast is a potent anti-inflammatory substance, a positive effect on this form of dermal disease is anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Patient (who is able to read, to write and to fully understand English language) has been informed both verbally and in writing about the objectives of the clinical study, the methods, the anticipated benefits and potential risks and the discomfort to which he/she may be exposed, and has given written consent to participation in the study prior to study start and any study-related procedure.
* Patient is suffering from mild to moderate plaque psoriasis
* Male or female patient of any ethnic origin, age 18 years or older presenting a minimum of 3% to a maximum of 10% BSA affected by mild to moderate plaque psoriasis proven by a dermatologist.
* Patient must have a minimum of 1 and a maximum of 3 in severity score of psoriasis
* Patient must have at least one target lesion of at least 1% BSA.
* Patient must be willing to wash out from current active therapy for at least 14 days prior to Day 1.
* Women of childbearing potential must have a negative pregnancy test at the Screening and Baseline Visits and agree to use a highly effective method of birth control. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner

Exclusion Criteria:

* Patient has spontaneously improving or rapidly deteriorating plaque psoriasis within at least the past 3 month.
* Patients who have a known history of psoriasis unresponsive to topical treatments.
* Patient has a physical condition (e.g., atopic dermatitis, contact dermatitis, tinea corporis) which, in the Investigator's opinion, might impair evaluation of plaque psoriasis or which exposes the patient to an unacceptable risk by trial participation.
* Clinically relevant abnormal laboratory values and vital signs suggesting an unknown underlying disease and requiring further clinical evaluation (as assessed by the Investigator).
* Patient is pregnant, nursing or planning a pregnancy during the trial period.
* Patient is currently enrolled in an investigational drug or device trial.
* Patient has received an investigational drug or an investigational device within 30 days prior to trial start.
* Patient has a history of allergic reactions to roflumilast or any inactive ingredients of the trial medication.
* Patient has positive results in any of the virology tests of acute or chronic infectious HIV and hepatitis virus infections.
* Abuse of alcohol or drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of clinical signs and symptoms score | 28 days

SECONDARY OUTCOMES:
Improvement of plaque psoriasis severity score, improvement of patient judged pruritus severity, change in dermal questionnaire, safety and efficacy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca